CLINICAL TRIAL: NCT02763670
Title: Comparison of Patient Care Management Strategies of Heart Failure in the Rhône-Alpes Region. A Clinical and Economic Study.
Brief Title: Patient Care Management Strategies for Severe Heart Failure in Rhône-Alpes, France.
Acronym: EFFICARD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2013.838
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2018-02

CONDITIONS: Severe Heart Failure
Keywords: Heart failure; patient education as topic; patient care management
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interventional (Other): PRETICARD patient care management
  Interventions: Other: PRETICARD patient care management
- Control (Other): Heterogenous "as usual" patient care management.
  Interventions: Other: "As usual " patient care management

INTERVENTIONS:
Other: PRETICARD patient care management — A standardized and specialized network to take care of the severe cardiac insufficiency:
  * An initial assessment and consultations with health professionals specialized in severe cardiac insufficiency during the hospitalization for cardiac insufficiency
  * At 1 months, consultations and acts realized by health professionals specialized (one hospital day care)
  * At 2 months, a therapeutic education program for heart failure patients, approved by the Rhône-Alpes regional public health authorities (week hospital: two days and one night).
  * At 6 and 18 months, one cardiology consultation
  * At 12 and 24 months, consultations and acts realized by health professionals specialized (one hospital day care)
  Arms: Interventional
Other: "As usual " patient care management — Conventional management of heart failure patients is defined in the guide HAS ("Haute Autorité de Santé") care course. Patient follow-up, however, is defined by the patient's physician and / or cardiologist at the waning of his hospitalization, according to the usual practice for patients with stage II, III or IV NYHA.
  According to these recommendations, the patient should see his cardiologist at least once a year.
  Usual practices are:
  * An initial assessment and consultations with health professionals specialized in severe cardiac insufficiency during the hospitalization for cardiac insufficiency
  * At 12 months, a cardiologic consultation. For the study, three evaluation points are programmed: two by phone at 6 and 18 months, two by a consultation at 24 months. This interview aimed to evaluate the number of hospitalization, consultations and acts realized by health professionals specialized (the information in the logbook).
  Arms: Control

SUMMARY:
The heart failure is a chronic pathology with prevalence from 2 to 3% of general population, a death rate of 50% at 6 months for patients with stage IV, and a probability of death or hospitalization or emergency consultation of 40% at 3 years. The care of patients is heterogeneous, especially in light of the organization of therapeutic education offered to patients and patient monitoring modalities.

The aim of this study is to investigate the management strategies for patients with chronic heart failure stage III or IV NYHA, and heart failure patients with stage II NYHA with previous hospitalization for heart failure.

This is a longitudinal observational multicenter study comparing a management strategy including patient education and monitoring as part of a hospital dedicated organization and an organization of care as usually done in France.

The primary endpoint was a composite endpoint of morbidity and mortality involving deaths, unplanned readmissions and emergency visits for heart failure.

The expected number of patients is 720 patients (360 per strategy). The follow-up duration of 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic heart failure patient with left ventricular ejection fraction (LVEF) defined by an impaired LVEF less than or equal to 40%.
* Heart failure stage III or IV NYHA, or heart failure patients with stage II NYHA with previous hospitalization for heart failure.
* Patient who has received a written or oral information of the study
* Patient affiliated with French health Insurance

Exclusion Criteria:

* Patient refusal to participate in the study
* Progressive neoplastic pathology.
* Patient with impaired cognitive functions known.
* Patient subject to a measure of socio-legal protection.
* Heart failure secondary to curable causes (an arrhythmia, valvular dysfunction, myocardial infarction, bypass surgery scheduled, aortic stenosis, breaking rope…)
* Dyspnea pulmonary origin: pulmonary arterial hypertension pre-capillary origin catheterization, defined by a Pcap ≤15 mmHg.
* Patient who underwent ventricular mechanical assistance.
* Patient with acute breathlessness is explained by: a severe lung infection (CPT <60% of predicted, ventricular ejection fraction <60% predicted) or pulmonary embolism or respiratory failure with ambient air PaO2 (arterial oxygen pressure) below 60 mmHg or oxygen therapy.
* Dialysis patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Actual)
Dates: Start 2015-09; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Composite endpoint combining the proportion of patients who died, the proportion of hospitalization for heart failure as well as the proportion of emergency visits for heart failure. | 12 months

SECONDARY OUTCOMES:
Unplanned re hospitalization rate or emergency consultations for cardiac insufficiency. | At 6, 18 and 24 months
Quality of life. | 12 months
  MINNESOTA Questionnaire.
Satisfaction. | 3 months
  Semi-structured interviews.
Cost of medical care | 24 months
  Identification of expenditure:
  * Hospitalizations
  * Consultations (inpatient and outpatient)
  * Biology and imaging
  * Medical transport

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: No